CLINICAL TRIAL: NCT02348138
Title: Effect of Isometric Handgrip Training on Cardiovascular Risk in Hypertensives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pernambuco (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Fundação de Amparo à Ciência e Tecnologia de Pernambuco (Other)
Responsible Party: Principal Investigator, Breno Quintella Farah, PhD student, University of Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISOPRESS
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Hypertension
Keywords: Isometric Handgrip
MeSH Terms: conditions — Hypertension | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Home-based isometric handgrip training (Experimental): All participants that will be assigned to home-based isometric handgrip training (HBT) will train three times per week for a total of 12 weeks, will perform a bout of isometric handgrip exercise: four sets of 2-min isometric contractions (using alternate hands) at 30% of maximal voluntary contraction; however, the training will be performed without daily supervision. Therefore, the subjects will receive a logbook to record the exercise sessions. In addition, visits will be scheduled at weeks 1, 3, 6, 9 and 11 to provide feedback to individuals and discuss potential problems in conducting training.
  Interventions: Other: Isometric handgrip training
- Supervised isometric handgrip training (Experimental): All participants that will be assigned to supervised isometric handgrip training (ST) will train three times per week for a total of 12 weeks, will perform a bout of isometric handgrip exercise: four sets of 2-min isometric contractions (using alternate hands) at 30% of maximal voluntary contraction with. The training will be performed with daily supervision.
  Interventions: Other: Isometric handgrip training
- Control group (No Intervention): Subjects randomized to the control group (CG) will be encouraged to increase the level of physical activity and make healthy eating, without, however, receive specific recommendations

INTERVENTIONS:
Other: Isometric handgrip training — The two experimental groups (HBT and ST) will receive intervention with isometric handgrip exercise for 12 weeks, and the HBT group without daily supervision.
  Other Names: Exercise
  Arms: Home-based isometric handgrip training; Supervised isometric handgrip training

SUMMARY:
The main purpose this study is to analyze the effects of isometric handgrip training on cardiovascular risk in hypertensive. For this, approximately 60 hypertensive, under anti-hypertensive medication, will be selected and randomly distributed into three groups: home-based isometric handgrip training (HBT), supervised isometric handgrip training (ST) and control group (CG).Subjects assigned to the HBT and ST will train three times per week for a total of 12 weeks, will perform a bout of isometric handgrip exercise: four sets of 2-min isometric contractions (using alternate hands) at 30% of maximal voluntary contraction. However, the subjects of the HBT group conduct the training without daily supervision. Subjects randomized to the CG will be encouraged to increase the level of physical activity and make healthy eating, without, however, receive specific recommendations.Baseline and after 12 weeks of intervention, the following cardiovascular risk indicators will be obtained: blood pressure, arterial stiffness, cardiac autonomic modulation, vasodilatory capacity and oxidative and inflammatory stress markers, in addition to microalbuminuria. For data analysis, in addition to descriptive statistics, two-way ANOVA for mixed model will be applied for within and between groups comparison. If the premises of this test are met. The level of significance that will be adopted is p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertension;
* Must be under anti-hypertensive medications of three months or more;
* May not present diabetes or other cardiovascular diseases;
* May not engaged in regular physical activity;
* May not have disabilities that compromise the physical activity practices.

Exclusion Criteria:

* Not perform more than 85% of the training sessions;
* Present diagnosis of metabolic diseases, cardiovascular or pulmonary during the study;
* Adherence to other physical activity program beyond the training offered by this study;
* Change in class and / or dose of medication during the study;
* Not using the medication regularly;
* Worsening of the disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in office blood pressure | Baseline and 12 weeks

SECONDARY OUTCOMES:
Change in ambulatory blood pressure | Basaline and 12 weeks
Change in central blood pressure | Basaline and 12 weeks
Change in cardiac autonomic modulation | Baseline and 12 weeks
Change in vasodilatory capacity | Baseline and 12 weeks
Change in arterial stiffness | Baseline and 12 weeks
Change in markers of oxidative stress | Baseline and 12 weeks
Change in markers of inflammation | Baseline and 12 weeks

OTHER OUTCOMES:
Adherence to training | 12 weeks
  Adherence to training will be evaluated by the number of subjects who completed the two types of training
Change in handgrip strength | Baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raphael M Ritti-Dias, Doctor, Study Director — University of Pernambuco; Breno Q Farah, Phd student, Principal Investigator — University of Pernambuco
Locations (1):
- University of Pernambuco, Recife, Pernambuco, Brazil